CLINICAL TRIAL: NCT05406960
Title: The Therapeutic Effect of Traditional Herbal Tea Infusion on Abnormal Uterine Bleeding- Menometrorrhagia
Brief Title: Therapeutic Effect of Herbal Infusion on Menometrorrhagia
Acronym: HERBALTREAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty of Medicine, Sousse (Other)
Collaborators: Centre Hôpital Universitaire Farhat Hached (Other)
Responsible Party: Principal Investigator, Pr. Hedi Khairi, Professor, dean of faculty, Faculty of Medicine, Sousse
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMSELMI
Record Dates: First submitted 2021-12-24; First posted 2022-06-07 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Abnormal Uterine Bleeding; Menorrhagia; Postmenopausal; Metrorrhagia; Hysterectomy; Heavy Menstrual Bleeding
Keywords: plants; Traditional herbal Medicine; Tisane
MeSH Terms: conditions — Metrorrhagia; Menorrhagia

STUDY DESIGN:
Intervention Model Description: The gynecologist who decided if the participant met the selection criteria or not Participants meeting the selection criteria will be included in the study.
  * Before starting all the included participants underwent a complete physical examination. Written informed consent will be obtained.
  * The herbal tea infusion will be self-administrated by participants at home.
  * Participants will receive training on how to make herbal tea infusions at home.
  * Participants will be interviewed by the investigator of the study:
  * To complete a quality-of-life questionnaire to determine the impact of the illness on their daily life.
  * Pictorial Bleeding Assessment Chart (PBAC): The history of the last menstruation period
  Participants will be asked to perform before starting the treatment :
  * Complete blood count (CBC)
  * Prothrombin Time (PT)
  * Prothrombin ratio (INR)
  * Fibrinogen (FIB) to detect bleeding disorders
  * serum Creatinine to detect urinary toxicity
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tea infusion (Experimental): The aerial parts of each plant were dried, then, they were powdered in a rotating knife grinder. The herbs were taken as tea infusion by the oral route. the powder of the mixture was added to 100 ml of boiling water and the tea infusion was taken three times a day for three consecutive days and it was repeated for three consecutive months
  Interventions: Dietary Supplement: Tea infusion

INTERVENTIONS:
Dietary Supplement: Tea infusion — Herbal tea infusion will be administrated by the oral route before food

SUMMARY:
This is an interventional, non-randomized, controlled, pilot study that explores a new approach to treat, Abnormal uterine bleeding-menometrorrhagia in women, being candidates for hysterectomy, based on tea infusion consumption of a mixture of two plants.

DETAILED DESCRIPTION:
Menometrorrhagia is excessive uterine bleeding resulting from a combination of two different conditions, namely menorrhagia, which is heavy bleeding during the menstrual period, and metrorrhagia, when the period lasts more than seven days or when uterine bleeding exists between periods. It is defined as abnormal uterine bleeding (AUB) and it is a worldwide health problem affecting 11 to 13% of the general female population in the reproductive age and increasing up to 24% in women aged 40-50 years. Conventional treatment of menometrorrhagia consists of symptomatic treatment including tranexamic acid and levonorgestrel intrauterine device. If the first-line medication fails to treat women with AUB, surgical treatment such as a hysterectomy could be necessary. However, both medical treatments and surgical procedures have different side effects, including gastrointestinal symptoms, liver disease, obesity, and thromboembolic diseases. Moreover, the hypoestrogenic state of these therapies can also lead to rapid bone demineralization and menopausal symptoms, such as vaginal dryness and hot flushes, having a negative effect on women's quality of life. Thus, because of these serious side effects, it seems logical to investigate other available sources. Such problems may be beyond the scope of herbal treatment.

Mentha pulegium is a perennial plant from the Lamiaceae family, also known as Pennyroyal, and is used in pharmaceutical and agro-alimentary industries. Artemisia abrotanum L, commonly known as Southernwood, is a small bushy shrub with small, feathery, narrow, and grey-green leaves. The genus belongs to the Asteraceae family.

A mixture of these two herbs is known as a strong emmenagogue.

Data collection:

The plants used in this study were collected through an ethnobotanical survey. The data on the plants' studies were collected through an internet search in: Medicinal plants mentioned in Canon www., www. Science Direct, www.pubmed.com. , www. Scopus, www.wiley.com, www. Google scholar, www. web of science, books in phytotherapy

All details with regard to :

* The effect of the treatment on the menstrual cycle
* Menstruation duration
* Adverse effects
* Bleeding intensity measured using Pictorial Blood Assessment Chart during three consecutive menstrual treatments and the three-month follow-up.

will be collected from participants by phone

Details about the Follow-up:

Allocated to intervention :

Follow-up (Visit 2): Phone or direct contact after the end of oral administration (day 3) for clinical response evaluation.

Phone or direct contact one week after treatment Follow-up 3: Phone or direct contact after the end of oral administration (day 3) for clinical response evaluation.

Phone or direct contact one week after treatment Follow-up (Visit 4): Phone or direct contact after the end of oral administration (day 3) for clinical response evaluation.

Phone or direct contact one week after treatment VISIT 5 (closing visit)

Statistical Analysis

Data entry and analysis will be performed using ( IBMV SPSS R 20.0). To test for normality and distribution of the variables. A significance level of a p-value of less than 0.05 will be considered Descriptive statistics will be used to examine the characteristics of the study population (means, standard deviation).

Comparison of the biological parameters and scores of PBAC between baseline and the end of treatment will be performed using paired t-test when variables are normally distributed and Wilcoxon signed ranks test, as a non-parametric test when variables are not normally distributed.

Sample size

The sample size will be assessed according to the following formula N = (Zα/2) 2 s2 /d2, where "s" is the standard deviation (SD ).

"d" is the accuracy of the estimate. "Zα/2" is the normal deviate for a two-tailed alternative hypothesis at a level of significance.

ELIGIBILITY:
Inclusion Criteria:

* Women failed first-line intervention to stop bleeding and planned for hysterectomy
* Women between (30-50 years)
* Able to understand and provide informed consent to participate in the study.
* Not pregnant or lactating
* Having menstrual period more than 7 days with uterine bleeding at irregular intervals.

Exclusion Criteria:

Participants with at least one of the following criteria will not be included in the trial:

* Chronic disease with long-term treatment (i.e. asthma, cardiovascular disorders..)
* woman taking any standard medications for abnormal uterine bleeding
* Women who have a history of gastrointestinal bleeding or ulcer
* Women who have abnormal kidney function
* Participants with increasing menstrual bleeding during the treatment requires surgical emergency procedures.
* Those refusing the instructions or participating in other clinical trials.
* Participant take other herbal treatment
* - Age less than 18 years
* - Healthy Volunteers
* women with ovarian tumours

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women suffering from AUB and being candidates for hysterectomy
Enrollment: 13 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2021-02-10 (Actual)

PRIMARY OUTCOMES:
Reduce the menstrual duration in days | 180 days
  the Pictorial Blood Loss Assessment Chart (PBLAC) the number of bleeding day during menstruation
Reduce the bleeding abundance | 180 days
  bleeding abundance will be measured by the Pictorial Blood Loss Assessment Chart (PBLAC) The total score is calculated by adding up the sum of all scores for the sanitary pads used in the menstrual cycle. : 1 for lightly stained, 5 for moderately soiled, and 20 for completely saturated pads. Clots were given a score of 1 for small and 5 for large clots.
  Abnormal PBLAC bleeding score greater than or equal to 100, which correlates with bleeding abundance, defined as greater than 80 mL of menstrual blood loss. Normal bleeding is defined as a score of 75 or less. A score of 0 indicates amenorrhea or the absence of menstruation.

SECONDARY OUTCOMES:
Change From Baseline in Hematocrit (Hct) Concentrations at Treatment Day 90 | 180 days
  Hematocrit was measured before treatment and after 90 days at the end of treatment
Change From Baseline in Hemoglobin Concentration at Treatment Day 90 | 90 days
  Hemoglobin was measured before treatment and after 90 day A positive value indicates an increase in hemoglobin from baseline at treatment day 90
Change From Baseline in Fibrinogen Concentration at Treatment Day 90 | 90 days
  Fibrinogen Concentration was measured before treatment and after 90 day
Change From Baseline in Prothrombin Time at Treatment Day 90 | 90 days
  Prothrombin Time was measured before treatment and after 90 day
hange From Baseline in serum Creatinine Time at Treatment Day 90 | 90 days
  to detect urinary toxicity. conducted at the start of the trial and after the last infusion consumption days 90

CONTACTS AND LOCATIONS:
Overall Officials: Hedi Khairi, Pr, Study Director — CHU, Farhat Hched Hospital, Faculty of medicine sousse tunisia 4000 Sousse Tunisia; Latifa Lassoued, Pr.Ag, Study Director — CHU Farhat Hached Hospital, Faculty of medicin Sousse,4000,Sousse,Tunisia
Locations (1):
- faculty of medicine Sousse, Sousse, Tunisia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Donnez J, Squifflet J, Donnez O. Minimally invasive gynecologic procedures. Curr Opin Obstet Gynecol. 2011 Aug;23(4):289-95. doi: 10.1097/GCO.0b013e328348a283. PMID 21666466
- [Background] Bone, K., and Mills, S. Principles and practice of phytotherapy: Modern Herbal Medicine. Churchill Livingstone.2nd ed. Londo n: Elsevier. 2013; 9780702052972
- [Background] Istre O, Langebrekke A, Qvigstad E. Changing hysterectomy technique from open abdominal to laparoscopic: new trend in Oslo, Norway. J Minim Invasive Gynecol. 2007 Jan-Feb;14(1):74-7. doi: 10.1016/j.jmig.2006.08.011. PMID 17218234
- [Background] Jazani NH, Ghasemnejad-Berenji H, Sadegpoor S. Antibacterial effects of Iranian Mentha pulegium essential oil on isolates of Klebsiella sp. Pak J Biol Sci. 2009 Jan 15;12(2):183-5. doi: 10.3923/pjbs.2009.183.185. PMID 19579942
- [Background] Kowalski R, Wawrzykowski J, Zawiślak G.Analysis of essential oils and extracts from Artemisia abrotanum L. and Artemisia dracunculus L. Herba Pol.2007.53: 246-254.
- [Background] Teri Moser Woo, Marylou Robinson.Pharmaco therapeutics for Advance Practice Nurse Prescribers. Library of Congress. (2016:138-1520.
- [Background] European Tea Committee (ETC), European Herbal Infusions Association (EHIA).Inventory List of Herbals Considered as Food. 2016 Available at: https://thie-online.eu/files/thie/docs/2019-09-26_PU_THIE_Inventory_List_status_27-06-2019_final.pdf
- [Background] Sutour S, Bradesi P, Casanova J, Tomi F. Composition and chemical variability of Mentha suaveolens ssp. suaveolens and M. suaveolens ssp. insularis from Corsica. Chem Biodivers. 2010 Apr;7(4):1002-8. doi: 10.1002/cbdv.200900365. PMID 20397217
- [Background] Fraser IS, Critchley HO, Munro MG, Broder M. Can we achieve international agreement on terminologies and definitions used to describe abnormalities of menstrual bleeding? Hum Reprod. 2007 Mar;22(3):635-43. doi: 10.1093/humrep/del478. Epub 2007 Jan 4. PMID 17204526
- [Background] Oueslati, S, Karray-Bouraoui, N, Attia, H. et al. Physiological and antioxidant responses of Mentha pulegium (Pennyroyal) to salt stress. Acta Physiol Plant 32. 2010.289-296. https://doi.org/10.1007/s11738-009-0406-0
- [Background] Chopra, R.N, Nayar S.L, Chopra, I.C. Glossary of Indian Medicinal Plant, New Delhi. CSIR.1956 .1-330.
- [Background] Hoffmann TC, Montori VM, Del Mar C. The connection between evidence-based medicine and shared decision making. JAMA. 2014 Oct 1;312(13):1295-6. doi: 10.1001/jama.2014.10186. No abstract available. PMID 25268434
- [Background] Qaraaty M, Kamali SH, Dabaghian FH, Zafarghandi N, Mokaberinejad R, Mobli M, Amin G, Naseri M, Kamalinejad M, Amin M, Ghaseminejad A, HosseiniKhabiri SJ, Talei D. Effect of myrtle fruit syrup on abnormal uterine bleeding: a randomized double-blind, placebo-controlled pilot study. Daru. 2014 Jun 2;22(1):45. doi: 10.1186/2008-2231-22-45. PMID 24888316
- [Background] Kang M, Ragan BG, Park JH. Issues in outcomes research: an overview of randomization techniques for clinical trials. J Athl Train. 2008 Apr-Jun;43(2):215-21. doi: 10.4085/1062-6050-43.2.215. PMID 18345348